CLINICAL TRIAL: NCT03361371
Title: Suctioning of NOse Therapy in Bronchiolitis - a Randomized Clinical Trial
Brief Title: Suctioning of NOse Therapy in Bronchiolitis
Acronym: SNOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Children's Hospital of Eastern Ontario (Other); London Health Sciences Centre (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Suzanne Schuh, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1671
Record Dates: First submitted 2017-11-21; First posted 2017-12-04 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Bronchiolitis
Keywords: Nose suctioning; Pediatric
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Prospective interventional.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional group (Experimental): Intervention Group: in addition to receiving the aforementioned bronchiolitis discharge instructions, this group will undergo nasal suctioning prior to each feeding as needed for 72 hours post discharge home, using exclusively the Zo-Li study device (see above under study device), with saline nose drops. Families in this group will be given the Zo-Li device at no cost and instructed in the appropriate technique and importance of using this tool.
  We shall not reveal the identity of the study devices to the ED physicians in order to minimize contamination of the control group. The ED treating physicians will also be blinded to which device the infant had been randomized to. We shall also ask the ED treating physicians not to recommend specific suctioning devices to the study patients.
  Interventions: Device: Battery operated nasal aspirator
- Control group (Placebo Comparator): Control Group: this group will receive standardized routine discharge instructions describing information about bronchiolitis, expected course of illness, recommended management strategies such as fever control, augmented air humidification, need for frequent feeding and warning signs prompting return for care. This group will be suctioned prior to feeds via bulb suction (with saline drops) which is expected to provide minimal effect, due to non-sustained negative pressures generated during bulb release. Since the benefit of nasal suction in bronchiolitis is unknown, this design is ethically reasonable. However, the use of no suction would likely meet with parental resistance and enrollment would be difficult. Families in the control group will be given the bulb device at no cost and instructed in the appropriate technique of using this tool prior to feeds.
  Interventions: Device: Suction bulb

INTERVENTIONS:
Device: Battery operated nasal aspirator — Suctioning prior to every feed with battery operated nasal aspirator for three days in addition to the routine standard of care.
  Arms: Interventional group
Device: Suction bulb — Suctioning prior to every feed with bulb nasal aspirator for three days in addition to the routine standard of care.
  Arms: Control group

SUMMARY:
Research Questions:

Primary:

In otherwise healthy infants 4 weeks to 12 months of age discharged home from the ED with acute bronchiolitis,1 is there a difference in the probability of "treatment failure" by 72 hours post discharge from the index ED visit in those receiving nasal suctioning via Zo-Li device prior to feeds compared to infants who receive nasal suctioning via bulb? Treatment failure is defined as 1) any bronchiolitis-related healthcare visit, except visits that have occurred only due to ED-recommendation at time of ED discharge or 2) the use of additional (non-study assigned) suctioning devices (see Outcome Measures section) within approximately 72 hours post discharge at the index ED visit.

Hypothesis:

We hypothesize that the infants who undergo scheduled nasal suctioning via ZoLi device will experience a lower treatment failure probability by approximately 72 hours post discharge from index ED visit compared to those managed by suction via a bulb.

Secondary:

1. In these infants, is there a difference in the mean number of medical visits for bronchiolitis (defined as #1 under primary outcome above) within 72 hours of ED discharge?
2. In these infants, is there a difference in the mean number of unscheduled medical visits for bronchiolitis within 72 hours of ED discharge?
3. In these infants, is there a difference in the mean number of ED visits for bronchiolitis within 72 hours of ED discharge?
4. In these infants, is there a difference in the probability of a parent reporting normal/near normal feeds on approximately 72 hours discharge?
5. In these infants, is there a difference in the probability of a parent reporting normal/near normal sleeping on approximately 72 hours post ED discharge?
6. For the parent, is there a difference in the probability of a parent reporting their own normal/near normal sleeping on approximately 72 hours post ED discharge?
7. In these infants, is there a difference in the probability of parents reporting at 72 hours post ED discharge as being "very satisfied" or "satisfied" with their ability to care for their child during the study period?

The sample size calculation is based on the assessment of the between-group difference in probability of treatment failure. The estimated total re-visit probability in bronchiolitis based on a recently published study was approximately 35% within 72 hours of ED discharge.49 In our pilot we have found the same rate of treatment failure. This is a superiority study in which the adoption of nasal suctioning will be recommended for future practice if the observed proportion of the primary outcome in this group is significantly lower than in the controls. With 162 patients per arm (324 in total) a two-sided test with a type I error of 0.05 will have 80% power to achieve statistical significance if suctioning reduces the probability of treatment failure from 40% to 25% (i.e. absolute reduction of 15%). This estimate is based on clinically relevant differences agreed upon by study investigators and it also represents an NNT of 7. In the Cochrane review of asthma therapies an NNT of a comparable magnitude led to a change in national practice recommendations.51 Since bronchiolitis and related medical visits are highly prevalent,20 this target difference would also have an important economic impact. Based on our previous bronchiolitis trials, the anticipated refusal rate may be 20%. Given the study design and our past experience, the study non-completion rate and loss to follow-up can safely be assumed to be no higher than 5% each. Therefore, to have complete data on 324 patients we plan to randomize 360 (i.e. 324/ (1 - 0.05) *(1 - 0.05) and to approach 450 (i.e. 360/ (1 - 0.20).

DETAILED DESCRIPTION:
This is a multi-center, randomized, outcome assessor- blinded clinical trial of infants discharged home from the ED with acute bronchiolitis. Two groups will be compared: infants receiving bronchiolitis suctioning via a bulb (see below) versus those given nasal suctioning via a battery-operated nasal aspiration Zo-Li device just prior to each feeding for 72 hours post index ED visit discharge. Evidence suggests that suctioning at frequent intervals is associated with movement of secretions from the lower airway with improved minute volume.40 The 72 hour study period has been chosen since the majority of infants discharged from the ED with bronchiolitis experience the targeted outcomes within this time frame.9

Prior to the ED discharge, all study participants will receive usual bronchiolitis care ordered by the ED physician as per standard of care which consists of supplemental oxygen for saturations <90% and supplemental IV hydration in those with inadequate oral intake.41 Eligible consenting patients deemed suitable for discharge home (representing approximately 60-70% of the bronchiolitis population presenting to the ED) will be randomly allocated to one of two study groups:

Control Group: this group will receive standardized routine discharge instructions describing information about bronchiolitis, expected course of illness, recommended management strategies such as fever control, augmented air humidification, need for frequent feeding and warning signs prompting return for care. This group will be suctioned prior to feeds via bulb suction (with saline drops) which is expected to provide minimal effect, due to non-sustained negative pressures generated during bulb release. Since the benefit of nasal suction in bronchiolitis is unknown, this design is ethically reasonable. However, the use of no suction would likely meet with parental resistance and enrollment would be difficult. Families in the control group will be given the bulb device at no cost and instructed in the appropriate technique of using this tool prior to feeds.

Intervention Group: in addition to receiving the aforementioned bronchiolitis discharge instructions, this group will undergo nasal suctioning prior to each feeding as needed for 72 hours post discharge home, using exclusively the Zo-Li study device (see above under study device), with saline nose drops. Families in this group will be given the Zo-Li device at no cost and instructed in the appropriate technique and importance of using this tool.

We shall not reveal the identity of the study devices to the ED physicians in order to minimize contamination of the control group. The ED treating physicians will also be blinded to which device the infant had been randomized to. We shall also ask the ED treating physicians not to recommend specific suctioning devices to the study patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of bronchiolitis in the ED as per the AAP diagnosis definition. Bronchiolitis is defined as the first episode of viral upper respiratory infection with respiratory distress and/or tachypnea for age.
2. Age 4 weeks up to and including 12 months of age. Participating infants will have to be at least 4 weeks post their expected due date of birth since infants with bronchiolitis below this age cut-off are at a much higher risk of apnea and dehydration than their older counterparts.
3. Nasal congestion as per parental report and/or the treating physician
4. Must have at least one of the following: home/cellular telephone or e- mail
5. Informed consent
6. Parent/Caregiver speaks English/French

Exclusion Criteria:

1. Previous diagnosis of bronchiolitis made more than 3 weeks prior to this ED visit.
2. Hospitalization at the index ED visit. Although we have considered starting the experimental intervention at presentation to the ED, this was deemed counterproductive since many patients with bronchiolitis are currently routinely suctioned in the ED which would likely contaminate the control arm and impact study results.
3. Use of any battery operated suctioning device prior to arrival. These families may choose to continue these electrical devices which would contaminate the study groups.

4- Co-morbidities which may impact outcomes such as known diagnosis of congenital heart disease, chronic respiratory disease including known lung disease due to prematurity, aspiration due to severe gastro-esophageal reflux, neuro-muscular/neurologic disease, immunodeficiency, coagulopathies, nasal/upper airway abnormalities, oral, gastrointestinal anomalies [except for corrected pyloric stenosis], tracheo-esophageal fistulas, gastric/gastro-jejunal tube feeding supplementation.

Ages: 4 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Treatment failure as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Occurrence of any of the following by day 3 post discharge home: Hospitalization for bronchiolitis, unscheduled medical visit, physician initiated visit for bronchiolitis within 3 days post discharge from initial ED visit

SECONDARY OUTCOMES:
Unscheduled, i.e. family-initiated return medical visit for bronchiolitis as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Family-initiated bronchiolitis-related medical visit
Emergency Department re-visit as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  ED visits for ongoing/worsening bronchiolitis symptoms
Feeding adequacy as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Normal/near normal feeding
Participant sleeping adequacy as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Normal/near normal sleeping pattern
Parental sleeping adequacy as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Normal/near normal sleeping pattern
Parental ability to care for their sick child as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Parental level of satisfaction for their ability to care for their child's illness

OTHER OUTCOMES:
Clinically important side-effects from nasal suctioning as measured by questionnaire administered on day 3 | Within 3 days post ED discharge at index visit
  Side-effects with the use of any suctioning device will be tracked

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Schuh, MD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

REFERENCES:
- [Derived] Schuh S, Coates AL, Sweeney J, Rumantir M, Eltorki M, Alqurashi W, Plint AC, Zemek R, Poonai N, Parkin PC, Soares D, Moineddin R, Finkelstein Y; Pediatric Emergency Research Canada (PERC) Network. Nasal Suctioning Therapy Among Infants With Bronchiolitis Discharged Home From the Emergency Department: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2337810. doi: 10.1001/jamanetworkopen.2023.37810. PMID 37856126